CLINICAL TRIAL: NCT06745414
Title: An Observational, Prospective and Retrospective Clinical Study to Evaluate the Performance of QIAstat-Dx® Gastrointestinal Panel 2 During Normal Conditions of Use
Brief Title: Clinical Performance of QIAstat-Dx® Gastrointestinal Panel 2
Status: Completed | Type: Observational
Sponsor: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: DHF-18-0129-0-CSP-001
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-01

CONDITIONS: Gastrointestinal Infection
Keywords: gastrointestinal infection; QIAstat-Dx; Clinical Performance Study

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fresh stool specimens in Cary-Blair transport media. Selected archived frozen stool specimens in Cary-Blair transport media will be tested retrospectively if required.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Performance evaluation of QIAstat-Dx® GI2 Panel using the QIAstat-Dx® Analyzer to demonstrate that the QIAstat-Dx® GI2 Panel achieves its intended performance during normal conditions of use by the intended user in the intended environment

DETAILED DESCRIPTION:
The objective of the study is to demonstrate that the QIAstat-Dx® Gastrointestinal Panel 2 achieves its intended performance during normal conditions of use by the intended user in the intended environment.

The primary objective is to evaluate the performance of QIAstat-Dx® GI2 Panel in comparison with the results obtained from the reference methods.

The secondary objective of the study is to evaluate the safety of QIAstat-Dx® GI2 Panel with respect to users/operators.

The primary study endpoint will be the results for each analyte obtained from testing prospective and retrospective specimens with QIAstat-Dx® GI2 Panel and Reference Method(s). Positive Percent Agreement (PPA) and Negative Percent Agreement (NPA) will be determined

ELIGIBILITY:
Inclusion Criteria:

1. Stool specimen must have been collected from subjects/patients which meet the institute's criteria for a suspected enteric pathogen, such as individuals presenting with symptoms of gastrointestinal infection;
2. Stool specimen will be residual and obtained for completion of routine gastrointestinal testing;
3. Specimen for testing will consist of stool specimens preserved in Cary- Blair medium following the manufacturer's instructions for use;
4. Fresh, unpreserved stool must be transferred to Cary-Blair as soon as possible after specimen collection;
5. When fresh stool is transferred into the Cary-Blair container, the maximum fill line of the container should not be exceeded;
6. There is an adequate residual volume (minimum 1.0 mL) of Cary- Blair preserved stool specimens;
7. Cary- Blair preserved stool specimens should represent a homogenous suspension (easily vortexed);
8. Cary- Blair preserved stool specimens have been stored at the following conditions prior testing:

   * Up to 4 days at Room Temperature (15 to 25˚C).
   * Up to 4 days at 2 to 8˚C (refrigerated);
9. Samples should be tested on the QIAstat-Dx® system and the reference method FilmArray within 3 hours of each other.

Exclusion Criteria:

1. Whole stool specimen that had been frozen;
2. Specimen that had been centrifuged;
3. Lack of clear subject identification or label on residual stool specimen;
4. Obvious physical damage of residual stool specimen;
5. Repeated specimens from the same subject;
6. Specimens in preservative collection media other than Cary-Blair;
7. Specimen containing formalin or any other fixative;
8. Rectal swab specimens
9. Specimens not collected according to manufacturer's instructions (under-filled or overfilled specimens);
10. Specimen contaminated with urine or water;
11. Leaking container.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with signs and symptoms of gastrointestinal infection
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical sensitivity | 8 months
  Positive percent agreement PPA
Clinical specificity | 8 months
  Negative percent agreement NPA

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Johnson, Principal Investigator — Qiagen Manchester Limited
Locations (1):
- QIAGEN, Manchester, United Kingdom